CLINICAL TRIAL: NCT05622136
Title: Dose-escalation Strategy of Regorafenib in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Dose-escalation of Regorafenib in Advanced Hepatocellular Carcinoma
Acronym: STRAT-aHCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Gomes da Fonseca, Principal Investigator,, Instituto do Cancer do Estado de São Paulo
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP3005
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma
Keywords: Regorafenib; Hepatocellular carcinoma; Dose; Tolerability; Quality of life
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Regorafenib (Experimental): Cycles 1 and 2:
  * Week 1: 80mg/day
  * Week 2: 120mg/day
  * Week 3: 160mg/day
  * Week 4: off-treatment Cycles 3 on (up to treatment discontinuation)
  * Weeks 1 to 3: Maximum dose tolerated daily, defined as the highest dose at which the patient had no adverse events grade ≥3 by CTCAE version 5.0 during cycles 1 and 2.
  * Week 4: off treatment
  * Dose adjustments may be required. Appendix 11.1 guide dose adjustments. Individual decisions at the occurrence of particular adverse events may be discussed individually within the study team and investigators.
  Treatment will be administered until any of the following events occur:
  * Both radiological and clinical progression according to definition of mRECIST or clinical deterioration that prevents treatment continuation according to the judgment of the attending physician
  * Limiting toxicity as defined by a grade 3 adverse event that does not resolve to grade < 3 within 7 days; adverse event grade 4 or 5.
  * Subject decision.
  Interventions: Drug: Regorafenib Oral Product

INTERVENTIONS:
Drug: Regorafenib Oral Product — Dose escalation strategy

SUMMARY:
The present protocol (STRAT-aHCC trial) aims to prospectively evaluate the tolerability, quality of life and efficacy of an alternative regimen of regorafenib in patients with advanced hepatocellular carcinoma (HCC) after progression to first-line. Patients will receive increasing dose of regorafenib in the first 2 treatment cycles (initial dose of 80mg, with weekly increments of 40mg up to 160mg in the first 2 treatment cycles). From the 3rd cycle on, the maximum tolerated dose during the first 2 cycles will be maintained. The maximum tolerated dose will be considered the highest dose in which the patient does not present grade ≥3 adverse events. The primary endpoint is the proportion of evaluable patients completing cycle 4. Radiologic response rate, quality of life, time to progression and overall survival will be evaluated as secondary endpoints.

DETAILED DESCRIPTION:
In patients who are refractory to first-line treatment with sorafenib, regorafenib was tested in the phase III RESORCE study. In this study, a standard dose of 160mg/day was used (in cycles of 4 weeks, with 3 weeks on treatment and 1 week off) until tumor progression or limiting toxicity. Regorafenib was superior to placebo with a significant increase in overall survival and became a sequential treatment option.

However, regorafenib is associated with relevant adverse events such as fatigue, hand-foot reaction, diarrhea and hypertension. Such events are more frequent in the first 2 cycles. In the RESORCE trial, 54% of patients had adverse events requiring interruption or dose reduction, and treatment discontinuation was required in 10% of patients. This toxicity profile limits the wide adoption of this drug in clinical practice.

Dose escalation strategies for regorafenib have been evaluated in patients with colorectal cancer and have resulted in better tolerability with comparable efficacy. However, there are no prospective studies with alternative doses of regorafenib in patients with advanced HCC.

The present protocol (STRAT-aHCC trial) aims to prospectively evaluate the tolerability, quality of life and efficacy of an alternative regimen of regorafenib in patients with advanced HCC. Patients will receive increasing dose of regorafenib in the first 2 treatment cycles (initial dose of 80mg, with weekly increments of 40mg up to 160mg in the first 2 treatment cycles - Figure 1). From the 3rd cycle on, the maximum tolerated dose during the first 2 cycles will be maintained. The maximum tolerated dose will be considered the highest dose in which the patient does not present grade ≥3 adverse events. The primary endpoint is the proportion of evaluable patients completing cycle 4. Radiologic response rate, quality of life, time to progression and overall survival will be evaluated as secondary endpoints.

Medical visits will be carried out weekly in the first 2 treatment cycles and every 4 weeks after the 3rd cycle. Laboratory tests will be performed every 2 weeks during the first 2 cycles and every 4 weeks after the 3rd cycle. Response assessment by imaging exams will be performed every 8 weeks. Quality of life assessments will be performed every 4 weeks using the EuroQol EQ-5D-5L7 questionnaire. The planned sample size is 28 patients with an expected duration of 25-30 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Hepatocellular carcinoma with histological or cytological confirmation or that meet radiological criteria for the diagnosis of HCC21;
3. BCLC-B stage not candidate for locoregional treatment or BCLC-C;
4. Have been previously treated with at least 1 line of systemic treatment with sorafenib, levantinib, atezolizumab plus bevacizumab or other immunotherapy-based regimen;
5. Have received the last dose of first-line systemic treatment between 2 and 6 weeks before starting study treatment;
6. Recovery to baseline or ≤ grade 1 from toxicities related to any previous treatments, unless the adverse event is not clinically significant as determined by the investigator (according to the Common Terminology Criteria for Adverse Events (CTCAE) v522);
7. Not having received previous treatment with regorafenib;
8. Child-Pugh A or B7 (in the absence of clinical ascites);
9. Measurable disease as defined by the RECIST 1.1 criteria. Target lesions must not have undergone previous local or locoregional treatment (example: ablation, transarterial chemoembolization, radiotherapy or selective internal radiotherapy)
10. Performance status: ECOG 0 or 1.
11. Adequate hematologic, hepatic and renal functions as defined below:

    i. Hemoglobin ≥ 8.5 g/dl ii. Absolute neutrophil count ≥ 1,000 /mm3 iii. Platelet count ≥ 50,000 /mm3 iv. Total bilirubin < 2.0 x upper limit of normality (ULN) v. ALT or AST <5 x LSN vi. Creatinine clearance (CrCI) ≥ 30 mL/min (according to Cockroft-Gault formula) vii. Serum albumin ≥ 2.8 mg/dl
12. Ability to understand informed consent and comply with the treatment protocol.
13. Informed consent form and clarification signed by the patient, impartial witness or legal representative.
14. Sexually active patients of childbearing potential and their partners must agree to use highly effective methods of contraception that result in a rate of less than 1% per year when used consistently and correctly throughout the study and 6 months after treatment discontinuation;
15. Female participants of childbearing potential cannot be pregnant at screening.

Exclusion Criteria:

1. Fibrolamellar carcinoma, sarcomatoid HCC or mixed hepatocellular cholangiocarcinoma;
2. Previous use of regorafenib;
3. Hepatic encephalopathy or medication requirement to control hepatic encephalopathy in the last 60 days before randomization;
4. Clinically significant ascites (ie, ascites that requires parcentesis or increased dose of diuretics) within 30 days prior to randomization.
5. Patients who have received local therapies (ablation, transarterial chemomebolization or surgery) within 28 days prior to randomization. Radiation treatments with the aim of pain control of bone metastases are allowed.
6. Known or suspected brain metastasis or cranial epidural disease unless adequately treated with surgery or radiotherapy and stable for at least 8 weeks from randomization.
7. Any participant who cannot be submitted neither to computed tomography (CT) nor magnetic resonance imaging (MRI) due to contra-indication to contrast media used.
8. The participant has an uncontrolled disease, or a significant complication in the last 28 days of randomization, such as:

   1. Cardiovascular disorders:

      * i. Class III or IV congestive heart failure as defined by the New York Heart Association, unstable angina pectoris, or symptomatic arrhythmias;
      * ii. Uncontrolled hypertension (defined as systolic blood pressure greater than 160 mmgHg or diastolic pressure > 95 mmHg despite antihypertensive therapy);
      * iii. Stroke, myocardial ischemia, or any ischemic event within the 6-month period prior to randomization;
   2. Gastrointestinal disorders, including those associated with a high risk of perforation:

      * i: active peptic ulcer disease, inflammatory bowel disease, tumors invading the gastrointestinal tract, diverticulitis, cholecystitis, appendicitis, acute pancreatitis and cholangitis;
      * ii: Abdominal fistula, gastro-intestinal perforation or abdominal abscess in the last 6 months;
      * iii: Esophageal varices that have not been adequately treated or that have been incompletely treated with bleeding or high risk of bleeding. Participants treated with adequate endoscopic therapy with no bleeding in the past 6 months are eligible;
   3. Clinically detected hematuria, hematemesis, melena, hemoptysis (>2.5 ml) or other clinically significant bleeding within the last 3 months of randomization.
   4. Cavitating pulmonary lesion or known manifestation of endobronchial disease;
   5. Other clinically significant diseases, at the discretion of the attending physician.
9. Majority surgery within 28 days of randomization. Minor surgeries within 10 days of randomization. Participants must have complete healing of the procedures prior to randomization;
10. History of psychiatric illness that is likely to interfere with the ability to understand the study procedures;
11. Pregnant or breastfeeding women;
12. Inability to swallow pills;
13. Known allergies to study drug components;
14. Any other known malignancy active at the time of randomization or diagnosis of another malignancy within two years of randomization, except superficial skin carcinomas or low-grade localized tumors considered cured and not treated with systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who complete 4 cycles of treatment | 4 months

SECONDARY OUTCOMES:
Proportion of patients with disease control after 4 treatment cycles; | 4 months
  Patients with partial response or stable disease after 4 cycles
Median overall survival: time from treatment initiation to death; | 5 years
  Time from treatment initiation to death
Median progression-free survival: time from treatment initiation to progression or death | 5 years
  Time from treatment initiation to progression or death
Score in the The 5-level EuroQol EQ-5D-5L questionnaire | 5 years
  - 0.532 (worst health state) and 1 (most optimal health state)

CONTACTS AND LOCATIONS:
Locations (1):
- ICESP - Instituto do Câncer do Estado de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No